CLINICAL TRIAL: NCT04290637
Title: The Galway Sea Swimmers Study: A Randomized Study of the Effect of Cold-Water Sea Swimming on Cardiovascular Risk Factors
Brief Title: The Galway Sea Swimmers Study
Acronym: GS3
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit during COVID-19 crisis
Sponsor: National University of Ireland, Galway, Ireland (Other)
Responsible Party: Principal Investigator, Prof. John William McEvoy, Professor, Preventive Cardiology, National University of Ireland, Galway, Ireland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C.A. 2327
Record Dates: First submitted 2020-02-24; First posted 2020-03-02 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-04

CONDITIONS: Cardiovascular Diseases; Hypertension
Keywords: Cardiovascular Diseases; Cardiac Disease; Heart Diseases; Hypertension; Blood Pressure; Swimming; Exercise; Vascular Stiffness; Pulse Wave Analysis; Health-Related Quality Of Life; Heart Rate Variability; Immersion
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Heart Diseases; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No sea swimming (Experimental): Stop sea swimming for 4-6 weeks
  Interventions: Other: No cold-water sea swimming
- Sea swimming (Active Comparator): Continue sea swimming for 4-6 weeks
  Interventions: Other: Cold-water sea swimming

INTERVENTIONS:
Other: Cold-water sea swimming — Continue sea swimming for 4-6 weeks
  Arms: Sea swimming
Other: No cold-water sea swimming — Discontinue sea swimming for 4-6 weeks
  Arms: No sea swimming

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of death worldwide. Hypertension is a well-established risk factor for the development of CVD. Lifestyle modifications, including exercise, remain the cornerstone of blood pressure (BP)-lowering strategy. Swimming has long been a popular recreational activity for exercise, and is recently gaining widespread recognition as an effective option in maintaining and improving cardiovascular health. Previous studies that involved pool swimming as an intervention (versus no pool swimming) demonstrated favorable benefits of the former on BP reduction. However, no studies to date have specifically investigated the effect of cold-water sea swimming on BP. Indeed, the naturally lower water temperature in the sea may engender a 'cold water immersion' experience in sea swimmers with subsequent stress physiology, which have been shown to exert unique effects on cardiovascular hemodynamics. This study primarily aims to determine the impact of cold-water sea swimming on BP in a group of habitual sea swimmers in Galway who will be randomly assigned to either continue or stop swimming for 4-6 weeks. Other objective and subjective health benefits to sea swimming will also be explored in this study. Given the ubiquitous nature of this activity in the Irish general public, particularly in Galway, this study has potential from a public health perspective, and would add to the literature base pertaining to the benefits of sea swimming on cardiovascular health.

DETAILED DESCRIPTION:
Consenting participants will be randomly assigned, 1:1, to either continuation of sea swimming or discontinuation of sea swimming for 4-6 weeks, stratified by the type of swimmer (those who purely immerse in the water for a brief period of time versus those who actually swim [i.e., exercise] in the water) and use of blood pressure medication at the time of study commencement (yes or no), using a block size of four to maintain balance between intervention arms. In line with previous studies that assessed the impact of swimming intervention on BP, participants randomized to the swimming arm should pursue sea swimming 2 or more days/week.

ELIGIBILITY:
Inclusion Criteria:

* habitual swimmers (i.e., sea swimming at least 2 times/week for the past year)
* 18 years of age or older
* able to provide informed consent

Exclusion Criteria:

* underlying cardiac (e.g., self-reported heart failure) or pulmonary diseases (e.g., self-reported chronic obstructive pulmonary disease)
* recent orthopedic procedures (e.g., joint replacement therapy)
* severe disabling comorbidity
* recent arm (both arms) or chest wall injury
* pregnant or breast feeding

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Change in mean systolic blood pressure | Measured at baseline and again at 6 weeks
  Systolic blood pressure recorded using a 24-hour ambulatory blood pressure monitor

SECONDARY OUTCOMES:
Change in Pulse Wave Velocity | Measured at baseline and 6 weeks
  Pulse wave velocity measured using Complior Device
Change in Augmentation index | Measured at baseline and 6 weeks
  Augmentation index measured using Complior device
Change in Heart rate variability | Measured at baseline and 6 weeks
  Measured using 24-hour ambulatory blood pressure monitor
Change in Health-related quality of life | Administered at baseline and 6 weeks
  Measure using EQ-VAS (visual analog scale) instrument. Values between 0 (worst imaginable health) and 100 (best imaginable health)
Change in mean diastolic blood pressure | Measured at baseline and again at 6 weeks
  Diastolic blood pressure recorded using a 24-hour ambulatory blood pressure monitor

OTHER OUTCOMES:
Change in Sleep quality | Administered at baseline and 6 weeks
  Measured using Pittsburgh Sleep Quality Index. Values between 0 and 21, higher score indicates worse sleep quality
Change in Muscular strength | Measured at baseline and 6 weeks
  Measured using Hand grip dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: John William McEvoy, MBBCh MHS, Principal Investigator — National University of Ireland, Galway
Locations (1):
- Croi Heart and Stroke Centre, Galway, Ireland

IPD SHARING:
Plan to Share IPD: No